CLINICAL TRIAL: NCT03522103
Title: Marijuana Harm Reduction: Innovative Strategies for Developing New Knowledge
Brief Title: Cannabis Observational Study on Mood, Inflammation, and Cognition
Acronym: COSMIC
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2547
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Inflammation; Inflammatory Response; Mood; Cognitive Change
Keywords: Cannabis; Marijuana; Cognition
MeSH Terms: conditions — Inflammation; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (including DNA analysis) and gut microbiome samples (including microbial DNA analysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project examines the effects of cannabis on cognition and other domains of function and whether those effects are dependent upon the ratio of THC to CBD in the product. Current cannabis users are asked to stop using their typical product and to use cannabis containing different ratios of the cannabinoids THC and CBD. Participants complete baseline assessments including cognitive tasks, clinical measures, substance use history, and blood draw. Participants then acquire and use their study strain on their own, and after a period of use the mobile pharmacology laboratory goes to a location of their choosing. They complete cognitive, motor and blood-based assessments, then leave the mobile lab to use their study product one last time, returning to the mobile lab to complete cognitive, motor, and blood-based assessments immediately after use and one hour after use. A small subset of participants complete all of these procedures but use edible as opposed to flower-based products.

DETAILED DESCRIPTION:
Cannabis research can be dated back to the 1970's where standardized smoking of low potency cannabis in a laboratory setting has been the primary method used to understand the effects of the drug. The objective of this program is to use a naturalistic design to advance a more nuanced understanding of the potential outcomes associated with using different strains of marijuana. Researchers need to understand the effects of commonly used cannabis strains, as they are used in every day life. Commonly available strains of cannabis sold in dispensaries in Colorado have 3-5 times greater potency of cannabinoids, such as the psychoactive compound tetrahydrocannabinol (THC), than what has been used in laboratory settings. It is possible that laboratory based studies underestimate the effects of more potent strains that are widely available. Also, scientists have focused on the effects of THC while mostly ignoring other major cannabinoids (e.g. cannabidiol or CBD) and their synergistic relationship.

The objective of this study is to observe how different strains of marijuana, based off their unique cannabinoid content, can influence your mental and physical state in real time. This program will allow researchers to observe these effects immediately before and after cannabis use. A participant will use cannabis in the comfort of their home, and will walk out their front door and into a mobile lab that will be parked outside of their house. In this study, there is no need to smoke and drive.

Participation is this study involves one appointment at the laboratory facility in Boulder and one appointment in the mobile laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Have prior experience with edibles
* Have used marijuana in the past month. This includes any form of marijuana consumption including flower, oil, wax, tinctures and edibles
* Not using other drugs (cocaine, opiates, methamphetamine) in the past 60 days
* Light alcohol use

Exclusion Criteria:

* Currently using a strain with greater than 1% CBD or less than 18% THC
* A University of Colorado student or employee
* Heavy tobacco use
* Are currently pregnant
* In treatment for psychotic disorder, bipolar disorder or schizophrenia

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Blood Cannabinoid Concentration | Change over 3 time points over 5 days: Baseline (before 5 days of use), Pre-Administration (after 5 days of use but prior to acute use), and Post-Administration (after 5 days of use but 60 minutes after acute use).
  To test the hypothesis that a high delta-9-tetrahydrocannabinol (THC) strain of marijuana will be associated with greater blood levels of THC and greater harmful effects, we will measure the concentrations of the cannabinoid THC in blood (ng/ml).
Change in Inflammation: Circulating Levels of cytokines (panel of inflammatory markers) | Change over 3 time points over 5 days: Baseline (before 5 days of use), Pre-Administration (after 5 days of use but prior to acute use), and Post-Administration (after 5 days of use but 60 minutes after acute use).
  Change in inflammation from before to after cannabis use will be tested in relation to THC and CBD blood levels.
The Drug Effects Questionnaire (DEQ) | Change over 2 time points over 1 hour: Pre-Administration (after 5 days of use but prior to acute self-administration), and Post-Administration (after 5 days of use but 60 minutes after acute self-administration).
  The DEQ is a 5 items visual analog scale used to measure the strength of marijuana as well as the desirable effects (de Wit & Phillips, 2012).
The Addiction Research Center Inventory (ARCI) | Change over 2 time points over 1 hour: Pre-Administration (after 5 days of use but prior to acute self-administration), and Post-Administration (after 5 days of use but 60 minutes after acute self-administration).
  The ARCI (Martin, Sloan, Sapira, & Jasinski, 1971), including the ARCI-Marijuana (M) scale (Chait, Fischman, & Schuster, 1985) will be used to measure subjective effects of marijuana in addition to drug-induced euphoria, stimulant-like effects, intellectual efficiency and energy, sedation, dysphoria, and other somatic effects.
Profile of Mood States (POMS) | Change over 3 time points over 5 days: Baseline (before 5 days of use), Pre-Administration (after 5 days of use but prior to acute use), and Post-Administration (after 5 days of use but 60 minutes after acute use).
  The Profile of Mood States (POMS) will be used to collect baseline information on mood as well as information on mood changes throughout the study. (Johanson & Uhlenhuth, 1980; McNair, Lorr, & Droppleman, 1971)
Cognitive Impairment | Change over 3 time points over 5 days: Baseline (before 5 days of use), Pre-Administration (after 5 days of use but prior to acute use), and Post-Administration (after 5 days of use but 60 minutes after acute use).
  Co-outcomes testing multiple domains of thinking, memory, and perception (NIH Toolbox), including the Flanker Inhibitory Control and Attention Task, Pattern Comparison Processing Speed Test, the Picture Sequence Memory Test, the List Sorting Working Memory Test, and immediate and delayed recall via the International Shopping List Test (ISLT). Cognitive outcomes are measured in standard scores (e.g. Range of >70 to >140 (Mean of 100 and SD of 15) with higher scores indicating better performance) and can be averaged to reflect a standard score of overall cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Hutchison, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MY, Kramer EB, Gibson LP, Bidwell LC, Hutchison KE, Bryan AD. Investigating the Relationship Between Cannabis Expectancies and Anxiety, Depression, and Pain Responses After Acute Flower and Edible Cannabis Use. Cannabis Cannabinoid Res. 2025 Feb;10(1):71-80. doi: 10.1089/can.2023.0264. Epub 2024 Apr 12. PMID 38608236
- [Derived] Gibson LP, Mueller RL, Winiger EA, Klawitter J, Sempio C, Williams S, Bryan AD, Bidwell LC, Hutchison KE. Cannabinoid Exposure and Subjective Effects of THC and CBD in Edible Cannabis Products. Cannabis Cannabinoid Res. 2024 Feb;9(1):320-334. doi: 10.1089/can.2022.0020. Epub 2022 Nov 15. PMID 36378267
- [Derived] Karoly HC, Milburn MA, Brooks-Russell A, Brown M, Streufert J, Bryan AD, Lovrich NP, DeJong W, Cinnamon Bidwell L. Effects of High-Potency Cannabis on Psychomotor Performance in Frequent Cannabis Users. Cannabis Cannabinoid Res. 2022 Feb;7(1):107-115. doi: 10.1089/can.2020.0048. Epub 2020 Sep 10. PMID 33998859